CLINICAL TRIAL: NCT03349528
Title: A Double-Blind Placebo-Controlled Trial of a Probiotic Supplement to Prevent Relapse and Improve the Clinical Course After Hospitalization for Bipolar Depression
Brief Title: Probiotics to Prevent Relapse After Hospitalization for Bipolar Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sheppard Pratt Health System (Other)
Responsible Party: Principal Investigator, Faith Dickerson, Principal Investigator, Stanley Research Program, Sheppard Pratt Health System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMRI/SPHS: 2017-01
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Bipolar Depression
Keywords: bipolar disorder; bipolar depression; depressive episode; probiotic supplement; probiotics; relapse prevention; rehospitalization
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic Supplement (Experimental): The probiotic supplement will consist of capsules containing approximately 1 billion (1.0 x 10^9) colony forming units of the probiotic organisms, Lactobacillus rhamnosus LGG® (LGG®) and Bifidobacterium animalis subsp. lactis BB-12® (BB-12®). The capsule, which will be swallowed, is a size 3 opaque, hard, hypromellose capsule. Participants will be asked to take 1 capsule of the probiotic supplement with a meal or with a snack daily for 24 weeks.
  Interventions: Biological: Probiotic Supplement
- Inert Compound (Placebo Comparator): The inert compound placebo looks identical to the probiotic supplement, and participants will be instructed to swallow 1 capsule with a meal or with a snack daily for 24 weeks.
  Interventions: Biological: Inert Compound

INTERVENTIONS:
Biological: Probiotic Supplement — Probiotic supplement 1 tablet by mouth daily
  Other Names: Probio-Tec® BG-VCap-6.5
  Arms: Probiotic Supplement
Biological: Inert Compound — Probiotic identical placebo 1 tablet by mouth daily
  Arms: Inert Compound

SUMMARY:
The purpose of this study is to determine if taking a probiotic supplement versus a placebo will reduce relapse and improve the clinical course among participants who have been hospitalized for bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (inclusive)
* Capacity for written informed consent
* Currently (or within the last 3 weeks) admitted to a Sheppard Pratt inpatient or day hospital program for symptoms of a depressive episode and a diagnosis Bipolar Disorder I or II, most recent episode depressed per Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5), the diagnosis of which is confirmed with the Structured Clinical Interview for DSM-5 Disorders (SCID-5)
* Proficient in the English language
* Available to come to Sheppard Pratt Towson for study visits after hospital discharge

Exclusion Criteria:

* Depressive symptoms better accounted for by a diagnosis of Major Depressive Disorder, Schizoaffective disorder, Schizophrenia, or disorder(s) other than Bipolar Disorder I or II
* DSM-5 diagnosis of intellectual disability or comparable diagnosis determined by previous version of the DSM
* Substance- or medically-induced mood symptoms at time of Visit 1/Baseline visit
* DSM-5 diagnosis of a moderate or severe substance use disorder, except for caffeine or tobacco, within three months prior to the Visit 1/Baseline visit
* History of IV drug use
* Any clinically significant or poorly controlled medical disorder as determined by the principal investigator and/or the study physician (e.g., HIV infection or other immunodeficiency condition, uncontrolled diabetes, congestive heart failure)
* A serious medical condition that affects brain or cognitive functioning (e.g., epilepsy, serious head injury, concussion involving loss of consciousness, brain tumor, or other neurological disorder)
* Pregnant, planning to become pregnant, or breastfeeding during the study period
* Documented celiac disease
* Participated in any investigational drug trial in the 30 days prior to the Visit 1/Baseline visit
* Receipt of Electroconvulsive therapy (ECT) in the 30 days prior to the Visit 1/Baseline visit or planned ECT after hospital discharge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Time to Relapse | Weeks 0 - 24 of study participation
  Time to relapse defined as time until psychiatric rehospitalization during the study period

SECONDARY OUTCOMES:
New Mood Episodes | Weeks 0 - 24 of study participation
  Number of new mood episodes determined by Structured Clinical Interview for DSM-5 Disorders (SCID-5), an interview using criteria from the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
Brief Psychiatric Rating Scale | Weeks 0 - 24 of study participation
  The Brief Psychiatric Rating Scale (BPRS) will be used to measure the severity of psychiatric symptoms. The BPRS contains 24 items, each rated on a scale from 1 (not present) to 7 (very severe). Total scores range from 24 to 168, and high scores indicate increased symptomatology.
Young Mania Rating Scale | Weeks 0 - 24 of study participation
  The Young Mania Rating Scale (YMRS) will be used to measure mania-related symptoms. The YMRS contains 11 items, each rated either on a scale from 0 to 4 or a scale from 0 to 8. Total scores range from 0 to 60, and higher scores indicate increased mania-related symptomatology.
Montgomery-Åsberg Depression Rating Scale (MADRS) | Weeks 0 - 24 of study participation
  The Montgomery-Åsberg Depression Rating Scale (MADRS) will be used to measure depression-related symptoms. The MADRS contains 10 items, each rated on a scale from 0 (none or normal) to 6 (most severe). Total scores range from 0 to 60, and higher scores indicate increased depression-related symptomatology.
Hamilton Depression Rating Scale | Weeks 0 - 24 of study participation
  The Hamilton Depression Rating Scale (HAM-D) will be used to measure depression-related symptoms. The HAM-D contains 24 items, each rated either on a scale from 0 to 2 or on a scale from 0 to 4. Total scores range from 0 to 76, and higher scores indicate increased depression-related symptomatology.
Columbia-Suicide Severity Rating Scale | Weeks 0 - 24 of study participation
  The Columbia-Suicide Severity Rating Scale (C-SSRS) measures suicide attempts and ideation. The C-SSRS is a tool containing one section of items used for assessing the specific type and intensity of suicidal ideation and one section of items used to determine number and type of suicide attempts and actual or potential lethality of the most lethal suicide attempt. The number of items used depends upon participant responses, and higher ratings on specific items indicate either more attempts, more intense ideation, or more lethal behavior. The C-SSRS will be used to determine the occurrence of suicide attempts or ideation.

OTHER OUTCOMES:
Intestinal Inflammation | Baseline, Week 12, Week 24
  Levels of intestinal inflammation as measured by antibodies to casein, gliadin and saccharomyces cerevisiae as well as C-reactive protein (CRP) and cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Faith Dickerson, PhD, MPH, Principal Investigator — Sheppart Pratt Health System
Locations (1):
- Sheppart Pratt Health System, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, symptom, and cognitive data will be shared with the National Database for Clinical Trials Related to Mental Illness (NDCT). Access may be obtained through an approved application with the NDCT.